CLINICAL TRIAL: NCT03419234
Title: Cabazitaxel With Abiraterone Versus Abiraterone Alone Randomized Trial for Extensive Disease Following Docetaxel: The CHAARTED2 Trial
Brief Title: Abiraterone Acetate and Antiandrogen Therapy With or Without Cabazitaxel and Prednisone in Treating Patients With Metastatic, Castration-Resistant Prostate Cancer Previously Treated With Docetaxel
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA8153; NCI-2017-00389 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8153 (Other: ECOG-ACRIN Cancer Research Group); EA8153 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma in the Soft Tissue; Prostate Carcinoma Metastatic in the Bone; Stage IV Prostate Adenocarcinoma AJCC v7
Keywords: prostate cancer; Castration-Resistant Prostate Cancer; Cabazitaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Androgen Antagonists; cabazitaxel; XRP6258; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (abiraterone acetate, prednisone, cabazitaxel) (Experimental): Patients receive abiraterone acetate PO QD on days 1-21, prednisone PO BID on days 1-21. Courses of abiraterone acetate and prednisone repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients receive cabazitaxel IV over 1 hour on day 1, and treatment with cabazitaxel repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care antiandrogen therapy with either LHRH agonist or antagonist, or surgical castration with bilateral orchiectomy.
  Interventions: Drug: Abiraterone Acetate; Drug: Androgen deprivation therapy; Drug: Cabazitaxel; Drug: Prednisone
- Arm B (abiraterone acetate, prednisone) (Active Comparator): Patients receive abiraterone acetate and prednisone as in Arm A. Patients also receive standard of care antiandrogen therapy with either LHRH agonist or antagonist, or surgical castration with bilateral orchiectomy.
  Interventions: Drug: Abiraterone Acetate; Drug: Androgen deprivation therapy; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: Zytiga
Drug: Androgen deprivation therapy — Receive standard of care antiandrogen therapy with either LHRH agonist or antagonist or surgical castration with bilateral orchiectomy.
Drug: Cabazitaxel — Given IV
  Other Names: Jevtana; RPR-116258A; Taxoid XRP6258; XRP-6258
  Arms: Arm A (abiraterone acetate, prednisone, cabazitaxel)
Drug: Prednisone — Given PO
  Other Names: Deltasone; Orasone; Medicorten; Panasol-S; Liquid-Pred

SUMMARY:
This randomized phase II trial studies how well abiraterone acetate and antiandrogen therapy, with or without cabazitaxel and prednisone, work in treating patients with castration-resistant prostate cancer previously treated with docetaxel that has spread to other parts of the body. Androgens can cause the growth of prostate cancer cells. Hormone therapy using abiraterone acetate and antiandrogen therapy may fight prostate cancer by lowering and/or blocking the use of androgens by the tumor cells. Drugs used in chemotherapy, such as cabazitaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving abiraterone acetate and antiandrogen therapy with or without cabazitaxel and prednisone may help kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether the addition of 6 cycles of cabazitaxel to abiraterone acetate in patients with castration-resistant prostate cancer (CRPC) that have previously received docetaxel and androgen deprivation therapy (ADT) for hormone-sensitive prostate cancer (HSPC) can improve progression-free survival (PFS) compared to abiraterone acetate alone.

SECONDARY OBJECTIVES:

I. To assess whether the addition of 6 cycles of cabazitaxel to abiraterone acetate in patients with CRPC that have previously received docetaxel and ADT for HSPC can increase the percentage of change in prostate-specific antigen (PSA) from baseline to week 12 of treatment as well as the maximum decline in PSA that occurs at any point after treatment compared to abiraterone acetate alone.

II. To assess whether the addition of 6 cycles of cabazitaxel to abiraterone acetate in patients with CRPC that have previously received docetaxel for HSPC can prolong time to PSA progression compared to abiraterone acetate alone.

III. To assess whether the addition of 6 cycles of cabazitaxel to abiraterone acetate in patients with CRPC that have previously received docetaxel for HSPC can improve radiographic response (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) compared to abiraterone acetate alone.

IV. To assess whether the addition of 6 cycles of cabazitaxel to abiraterone acetate in patients with CRPC that have previously received docetaxel and ADT for HSPC can prolong the overall survival (OS) compared to abiraterone acetate alone.

V. To assess safety and tolerability of the combination of 6 cycles of cabazitaxel and abiraterone acetate.

TERTIARY OBJECTIVES:

I. To examine whether patients with circulating tumor cells (CTCs) positive for AR-V7 at baseline have a longer radiographic or clinical PFS to the combination of cabazitaxel and abiraterone acetate vs. abiraterone acetate alone.

II. To examine whether the addition of cabazitaxel to abiraterone acetate can change the AR-V7 status of patients who are positive at study entry.

III. To examine whether the addition of cabazitaxel to abiraterone acetate has any impact on future development of AR-V7 positivity at the time of disease progression.

IV. To assess if the changes in total tumor burden from baseline to week 12 as assessed with sodium fluoride (NaF) positron emission tomography (PET)/computed tomography (CT) will differ between two arms.

V. To correlate total tumor burden at the baseline as assessed with NaF PET/CT with the PFS.

VI. To correlate heterogeneity of response from baseline to week 12 as assessed with NaF PET/CT with the PFS.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive abiraterone acetate orally (PO) once daily (QD) on days 1-21, prednisone PO twice daily (BID) on days 1-21. Courses of abiraterone acetate and prednisone repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients receive cabazitaxel intravenously (IV) over 1 hour on day 1, and treatment with cabazitaxel repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care antiandrogen therapy with either luteinizing hormone-releasing hormone (LHRH) agonist or antagonist, or surgical castration with bilateral orchiectomy.

ARM B: Patients receive abiraterone acetate and prednisone as in Arm A. Patients also receive standard of care antiandrogen therapy with either LHRH agonist or antagonist, or surgical castration with bilateral orchiectomy.

After completion of study treatment, patients are followed up every 3 or 6 months and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer (adenocarcinoma of the prostate)
* Previous chemotherapy with at least 3 cycles of docetaxel for hormone-sensitive metastatic prostate cancer
* Metastatic disease as evidenced by the presence of soft tissue and/or bone metastases on imaging studies (CT/magnetic resonance imaging [MRI] of abdomen/pelvis, bone scintigraphy or NaF PET/CT)
* Ability to swallow abiraterone acetate tablets as a whole
* All patients must be receiving standard of care androgen deprivation treatment (surgical castration versus LHRH agonist or antagonist treatment); subjects receiving LHRH agonist or antagonist must continue treatment throughout the time on this study
* Patients must have castrate serum level of testosterone of < 50 ng/dL (< 1.73 nmol/L)
* Patients must have progressive disease while receiving androgen deprivation therapy defined by any one of the following as per the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria for PSA, measurable disease or non-measurable (bone) disease during treatment with ADT:

  * PSA: At least two consecutive rises in serum PSA, obtained at a minimum of 1-week intervals, with the final value >= 1.0 ng/mL, confirmed <=4 weeks prior to randomization
  * Measurable disease (by RECIST 1.1): > 20% increase in the sum of the longest diameters of all measurable lesions or the development of new measurable lesions; the short axis of a target lymph node must be more than 15 mm to be assessed for change in size
  * Non-measurable (bone) disease: The appearance of two or more new areas of uptake on bone scan (or NaF PET/CT) consistent with metastatic disease compared to previous imaging during castration therapy; the increased uptake of pre-existing lesions on bone scan will not be taken to constitute progression, and ambiguous results must be confirmed by other imaging modalities (e.g. X-ray, CT or MRI). Clinical decisions about response or progression will be based on CT and bone scans.
* Patients may or may not have been treated previously with a nonsteroidal antiandrogen, such as flutamide, bicalutamide or nilutamide; for patients previously treated with an antiandrogen, they must be off treatment for at least 4 weeks (for flutamide) or 6 weeks (for bicalutamide or nilutamide) prior to registration and must have shown PSA progression after discontinuing the anti-androgen
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Hemoglobin (HgB) >= 9.0 gr/dL
* Platelets >= 100,000/mm^3
* Creatinine < 2.0 mg/dL
* Patients must be informed of the experimental nature of the study and its potential risks, and must sign an Institutional Review Board (IRB)-approved written informed consent form indicating such an understanding
* Patients with resected or irradiated brain metastases or those treated with stereotactic radiation therapy are eligible to enroll, provided that they do not require treatment with steroids that exceeds 10 mg of prednisone daily or equivalent
* Sexually active males must use an accepted and effective method of double barrier contraception or abstain from sexual intercourse for the duration of their participation in the study and for 26 weeks after the last dose of study drug
* NaF PET/CT OPTIONAL SUB-STUDY ELIGIBILITY CRITERIA

  * Ability to lie still for imaging
  * Weight =< 300 lbs (pounds)
  * Metastatic disease confined predominantly to the bones

Exclusion Criteria:

* Any prior chemotherapy or androgen receptor (AR)-directed therapy for CRPC, (e.g. docetaxel, cabazitaxel, mitoxantrone, abiraterone acetate, ketoconazole, or enzalutamide); previous treatment with radium-223 or sipuleucel-T is allowed
* Pure small cell or other variant (non-adenocarcinoma) prostate cancer histology for which treatment with abiraterone would not be considered appropriate
* Patients may not be receiving other therapeutic investigational agents or be receiving concurrent anticancer therapy other than standard androgen deprivation therapy; concurrent treatment with agents to prevent skeletal-related events (such as zoledronic acid or denosumab) will be allowed as long as it was initiated prior to study entry or there are plans to initiate it after cycle 2 day 1.
* Any medical condition for which prednisone (corticosteroid) is contraindicated
* Total bilirubin > upper limit of normal (ULN) (NOTE: in subjects with Gilbert's syndrome, if total bilirubin is > ULN, measure direct and indirect bilirubin and if direct bilirubin is within normal range, subject may be eligible)
* Alanine (ALT) or aspartate (AST) aminotransferase > 1.5 x ULN
* Active infection requiring treatment with antibiotics
* History of adrenal insufficiency or hypoaldosteronism
* Myocardial infarction or arterial thrombotic event within 6 months of randomization, heart failure of New York Heart Association class II or higher, uncontrolled angina, severe uncontrolled ventricular arrhythmia
* External beam radiation therapy within 2 weeks of registration
* Prior history of allergic reactions to G-CSF
* Prior history of allergic reactions to docetaxel and/or to medications formulated with polysorbate 80
* History of active malignancy; patients with a history of cancer that has been adequately treated and are free of disease recurrence for 3 years or more are allowed to participate; patients with non-melanoma skin cancers or carcinoma in situ of the bladder that have been adequately excised are eligible to participate
* Life expectancy of < 12 months at screening
* Grade >= 2 neuropathy
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 100 mmHg). Patients with a history of hypertension are allowed to enroll provided blood pressure is controlled with anti-hypertensive treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2026-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Kyriakopoulos, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (672):
- United States (665):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Veteran's Administration Medical Center - New Orleans, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Bloomfield, Bloomfield, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Veteran's Affairs Medical Center - Saint Louis, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kenansville, Kenansville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Vidant Oncology-Richlands, Richlands, North Carolina
  - Marion L Shepard Cancer Center at Vidant Beaufort Hospital, Washington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Abington Memorial Hospital-Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Bon Secours Maryview Medical Center, Portsmouth, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on February 8, 2018 and closed to accrual on March 26, 2021, after accrual of 223 patients.
Period: Overall Study
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone)
Started | 111 | 112
Patients who received protocol therapy | 109 | 108
Patients who started protocol therapy and had both baseline PSA as well as 12-week PSA available | 100 | 93
Completed | 0 | 0
Not Completed | 111 | 112
Not completed — Disease progression | 37 | 36
Not completed — Adverse Event | 6 | 9
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Death | 5 | 1
Not completed — Alternative therapy | 4 | 2
Not completed — PSA progression | 8 | 10
Not completed — Rising PSA and bone issues | 3 | 2
Not completed — Clinical deterioration/clinical progression/symptomatic progression | 10 | 16
Not completed — Physician Decision | 12 | 11
Not completed — Second malignancy | 1 | 0
Not completed — Insurance status change/patient could not afford | 2 | 1
Not completed — Non-compliance | 1 | 3
Not completed — Mistakenly off treatment | 1 | 0
Not completed — Transition to hospice | 1 | 0
Not completed — Still on treatment | 9 | 8
Not completed — Never received protocol therapy | 2 | 4
Not completed — Other complicating disease | 0 | 1
Not completed — patient switched from prednisone to another steroid | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients were included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone) | Total
Number analyzed (Participants) | 111 | 112 | 223
Age, Continuous [Median (Full Range); unit: years] | 63 [42 to 79] | 66 [41 to 80] | 64 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 111 | 112 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 104 | 105 | 209
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 22 | 42
  White | 84 | 81 | 165
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from randomization to radiographic progression, symptomatic deterioration requiring discontinuation of treatment or death, whichever occurs first. Patients who died without documented radiographic progression or symptomatic deterioration and the death occurred more than 6.5 months after the date of last disease assessment were censored at the date of last disease assessment.
Time Frame: Assessed every 9 weeks for the first 18 weeks, then every 12 weeks until treatment discontinuation; if treatment discontinued prior to radiographic progression, then every 3 months until radiographic progression, up to 5 years
Population: All randomized patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone)
Number analyzed (Participants) | 111 | 112
months | 14.9 [9.9 to 18.6] | 9.9 [7.0 to 12.6]
Statistical Analysis 1: Comparison: Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) vs Arm B (Abiraterone Acetate, Prednisone); Test type: Superiority; p = 0.049, Log Rank; Stratified log rank test

2. Secondary Outcome: Percent Change in PSA From Baseline to 12 Weeks
Description: PSA was assessed at baseline and 12 weeks. Percent change in PSA from baseline to 12 weeks is calculated as follows:
  ((PSA at 12 weeks - baseline PSA)/baseline PSA) x 100
Time Frame: Assessed at baseline and 12 weeks
Population: Patients who started protocol therapy and had both baseline PSA as well as 12-week PSA available are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of change in PSA
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone)
Number analyzed (Participants) | 100 | 93
percentage of change in PSA | -87.5 [-94.9 to -52.1] | -65.9 [-91.3 to -16.1]

3. Secondary Outcome: Maximum Percent Change in PSA From Baseline While on Treatment
Description: Maximum percent change in PSA from baseline while on treatment was calculated as follows:
  ((PSA nadir while on treatment - baseline PSA)/baseline PSA) x 100
Time Frame: Assessed at baseline, every 3 weeks for 18 weeks, then every 6 weeks until treatment discontinuation, up to 5 years
Population: Patients who started protocol therapy are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of change in PSA
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone)
Number analyzed (Participants) | 109 | 108
percentage of change in PSA | -94.0 [-98.1 to -65.8] | -67.7 [-94.8 to -15.5]

4. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was defined as the time from randomization to PSA progression or date of last PSA assessment. Patients who experienced radiographic progression without documented PSA progression were counted as having an event.
Time Frame: Assessed at baseline, every 3 weeks for 18 weeks, then every 6 weeks until treatment discontinuation, up to 5 years
Population: All randomized patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone)
Number analyzed (Participants) | 111 | 112
months | 10.0 [8.5 to 13.5] | 6.1 [4.4 to 8.0]

5. Secondary Outcome: Proportion of Patients With Radiographic Response
Description: Radiographic response was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and was defined as either complete response (CR) or partial response (PR).
  CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. All (non-target) lymph nodes must be non-pathological in size (< 10 mm short axis).
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 1
Population: All randomized patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone)
Number analyzed (Participants) | 111 | 112
Proportion of participants | 0.117 [0.064 to 0.192] | 0.080 [0.037 to 0.147]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization until death or date last known alive.
Time Frame: Assessed every 3 month is patient is < 2 years from study entry, every 6 months if patient is 2-3 years from study entry, and then annually for up to year 5
Population: All randomized patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone)
Number analyzed (Participants) | 111 | 112
months | 25.0 [20.6 to 32.5] | 26.9 [19.6 to 29.4]

7. Other Pre Specified Outcome: PFS Among Patients With Circulating Tumor Cells (CTCs) Positive for Androgen-receptor Splice Variant 7 Messenger RNA (AR-V7) at Baseline
Description: PFS is defined as time from randomization to radiographic progression, symptomatic deterioration requiring discontinuation of treatment or death, whichever occurs first. Patients who died without documented radiographic progression or symptomatic deterioration and the death occurred more than 6.5 months after the date of last disease assessment were censored at the date of last disease assessment. AR-V7 was assessed at baseline.
Time Frame: Assessed at baseline, every 9 weeks for the first 18 weeks, then every 12 weeks until treatment discontinuation; if treatment discontinued prior to radiographic progression, then every 3 months until radiographic progression, up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Androgen-Receptor Splice Variant 7 Messenger RNA (AR-V7) Status
Description: The presence of AR-V7 in circulating tumor cells was assessed at baseline and Cycle 5 Day 1.
Time Frame: Assessed at baseline and Cycle 5 Day 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Development of AR-V7 Positivity at the Time of Disease Progression
Description: The presence of AR-V7 in circulating tumor cells was assessed at baseline and disease progression.
Time Frame: Assessed at baseline and disease progression
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Total Tumor Burden From Baseline to Week 12 as Assessed With NaF PET/CT
Description: Total tumor burden was assessed by NaF PET/CT at baseline and 12 weeks. The changes in total tumor burden will be compared between the two arms.
Time Frame: Assessed at baseline and 12 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Association Between PFS and Total Tumor Burden at the Baseline as Assessed With NaF PET/CT
Description: PFS is defined as time from randomization to radiographic progression, symptomatic deterioration requiring discontinuation of treatment or death, whichever occurs first. Patients who died without documented radiographic progression or symptomatic deterioration and the death occurred more than 6.5 months after the date of last disease assessment were censored at the date of last disease assessment. The association between PFS and total tumor burden at baseline as assessed with NaF PET/CT will be evaluated.
Time Frame: as for outcome 7
Reporting Status: Not Posted

12. Other Pre Specified Outcome: The Association Between PFS and the Heterogeneity of Response From Baseline to Week 12 as Assessed With NaF PET/CT
Description: PFS is defined as time from randomization to radiographic progression, symptomatic deterioration requiring discontinuation of treatment or death, whichever occurs first. Patients who died without documented radiographic progression or symptomatic deterioration and the death occurred more than 6.5 months after the date of last disease assessment were censored at the date of last disease assessment. The association between PFS and the heterogeneity of response from baseline to week 12 as assessed with NaF PET/CT will be evaluated.
Time Frame: Assessed at baseline, 12 weeks, every 9 weeks for the first 18 weeks, then every 12 weeks until treatment discontinuation; if treatment discontinued prior to radiographic progression, then every 3 months until radiographic progression, up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment, up to 5 years
Description: All randomized patients are included in the analysis of all-cause mortality. Only patients who received protocol therapy are included in the analysis of adverse events.
Arm/Group | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) | Arm B (Abiraterone Acetate, Prednisone)
All-Cause Mortality (participants affected / at risk) | 80/111 | 79/112
Serious Adverse Events (participants affected / at risk) | 46/109 | 31/108
Other Adverse Events (participants affected / at risk) | 101/109 | 80/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) (N=109) | Arm B (Abiraterone Acetate, Prednisone) (N=108)
Anemia (Blood and lymphatic system disorders) | 7 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Fatigue (General disorders and administration site conditions) | 6 | 2
Fever (General disorders and administration site conditions) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 5 | 0
Alanine aminotransferase increased (Investigations) | 1 | 5
Alkaline phosphatase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 4 | 2
Lymphocyte count increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 11 | 0
Platelet count decreased (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 9 | 0
Investigations - Other, specify (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 4 | 4
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 11 | 12
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Abiraterone Acetate, Prednisone, Cabazitaxel) (N=109) | Arm B (Abiraterone Acetate, Prednisone) (N=108)
Anemia (Blood and lymphatic system disorders) | 60 | 30
Edema limbs (General disorders and administration site conditions) | 22 | 13
Fatigue (General disorders and administration site conditions) | 78 | 47
Constipation (Gastrointestinal disorders) | 12 | 8
Diarrhea (Gastrointestinal disorders) | 37 | 6
Nausea (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 18 | 4
Urinary tract infection (Infections and infestations) | 7 | 2
Lymphocyte count decreased (Investigations) | 14 | 3
Neutrophil count decreased (Investigations) | 8 | 1
White blood cell decreased (Investigations) | 7 | 1
Anorexia (Metabolism and nutrition disorders) | 7 | 1
Hypokalemia (Metabolism and nutrition disorders) | 19 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Hypertension (Vascular disorders) | 37 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT03419234/Prot_SAP_000.pdf